CLINICAL TRIAL: NCT04829344
Title: A Randomized, Double-Masked, Vehicle-Controlled, Parallel Evaluation of the Local Anesthetic Effect of Articaine Sterile Topical Ophthalmic Solution
Brief Title: A Study of the Safety and Anesthetic Effect of AG-920 Topical Ophthalmic Solution
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Genomics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AG-920-CS302
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Anesthesia, Local
Keywords: AG-920; articaine; septocaine; Intravitreal Injection
MeSH Terms: interventions — Carticaine

STUDY DESIGN:
Intervention Model Description: Subjects who provide informed consent and fulfill all the inclusion criteria and none of the exclusion criteria will be randomized in a 1:1 ratio to receive a single dose of AG-920 or identical looking placebo into one (study) eye (2 drops 30 seconds apart).
Who Masked: Participant, Investigator
Masking Description: The Investigator(s), Sponsor, and the subject will be masked to treatment assignment throughout the conduct of the study. Exceptions to this are limited to one statistician at the Contract Research Organization (CRO) who will prepare the randomization code, and three people at the Sponsor who will review the batch records and release product. None of these unmasked persons will be involved in the day to day execution of the study. The masking will be broken after database lock.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AG-920 (Experimental): Articaine Sterile Topical Ophthalmic Solution (AG-920) is a sterile, isotonic, non-preserved aqueous solution containing the active ingredient Articaine HCl 8%, Boric Acid, Mannitol, Sodium Acetate Trihydrate, Glacial Acetic Acid, and Edetate Disodium Dihydrate. The product formulation is adjusted to pH 4.5 to 5.0. Each subject randomized to AG-920 will receive a single dose of 2 drops 30 seconds apart from a single vial into study eye.
  Interventions: Drug: AG-920
- Placebo (Placebo Comparator): Placebo ophthalmic solution is identical to the active product, with the exception of the active ingredient. Each subject randomized to placebo will receive a single dose of 2 drops 30 seconds apart from a single vial into study eye.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AG-920 — AG-920 Sterile Topical Ophthalmic Solution
  Other Names: articaine
  Arms: AG-920
Drug: Placebo — Placebo Topical Ophthalmic Solution
  Arms: Placebo

SUMMARY:
This is a Phase 3, randomized, placebo-controlled, double masked, parallel design study in healthy subjects performed in the US. It is designed to evaluate the safety and anesthetic efficacy of AG-920 Sterile Topical Ophthalmic Solution.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, placebo-controlled, double masked, parallel design study in healthy subjects performed in the US. It is designed to evaluate the safety and anesthetic efficacy of AG-920 Sterile Topical Ophthalmic Solution. In this study, subjects who provide informed consent and fulfill all the inclusion criteria and none of the exclusion criteria will be randomized in a 1:1 ratio to receive a single dose of AG-920 or identical looking placebo into the study eye. Subjects will undergo a conjunctival pinch procedure and the pain associated with the pinch rated.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to any study-related procedures being performed.
2. Is male or a non-pregnant, non-lactating female aged 18 years or older.
3. Willing and able to follow instructions and be present for the required study visits.
4. Have an Early Treatment Diabetic Retinopathy Study (ETDRS) Best Correct Visual Acuity (BCVA) of 20/200 or better in each eye.
5. Have an Intraocular Pressure (IOP) between 7 and 30 mmHg.
6. Certified as healthy by clinical assessment.
7. Verbal communication skills adequate to participate.
8. Able to tolerate bilateral instillation of Over-The-Counter artificial tear product based on investigator judgement.

Exclusion Criteria:

1. Have participated in an investigational study within the past 30 days.
2. Have a contraindication to local anesthetics.
3. Have known decreased corneal or conjunctival sensitivity.
4. Have had ocular surgery in either eye within the past 90 days.
5. Have had an intravitreal injection in either eye within 14 days.
6. Have ocular disease requiring punctual plugs or ocular inflammation.
7. Are currently using a systemic opioid or opiate analgesic or topical NSAID.
8. Cannot withhold their over the counter (OTC) artificial tear lubricant products for one hour preceding or following study medication.
9. Any condition, including alcohol or drug dependency, that would limit the subject's ability to comply with the procedures of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Uram, MD, Study Director — Medical Expert
Locations (1):
- American Genomics Site 2, McAllen, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez VH, Wirta DL, Uram M, Schupp A, Widmann M, Novack GD. Two Randomized, Double-masked, Placebo-controlled Studies of the Local Anesthetic Effect of Articaine Ophthalmic Solution. Clin Ophthalmol. 2023 May 10;17:1357-1365. doi: 10.2147/OPTH.S409241. eCollection 2023. PMID 37192994

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred and twenty one (121) subjects were screened, of which 120 were randomized and treated, all of whom completed the study. First subject screened 30March2021, last subject completed 10May2021.
Period: Overall Study
Arm/Group | AG-920 | Placebo
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AG-920 | Placebo | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 56 | 60 | 116
  >=65 years | 4 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: year] | 34.9 (15.6) | 37.0 (14.4) | 35.9 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 36 | 67
  Male | 29 | 24 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 59 | 59 | 118
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 58 | 58 | 116
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120
BCVA LogMar Study Eye [Mean (Standard Deviation); unit: LogMar] | 0.0 (0.1) | 0.0 (0.1) | 0.0 (0.1)
BCVA LogMar Fellow Eye [Mean (Standard Deviation); unit: LogMar] | 0.0 (0.1) | 0.0 (0.1) | 0.0 (0.1)
Color of Iris [Count of Participants; unit: Participants]
  Black | 0 | 2 | 2
  Brown | 56 | 50 | 106
  Green | 0 | 2 | 2
  Hazel | 4 | 6 | 10
IOP Study Eye [Mean (Standard Deviation); unit: mmHg] | 14.6 (2.7) | 14.5 (2.6) | 14.5 (2.6)
IOP Fellow Eye [Mean (Standard Deviation); unit: mmHg] | 14.7 (2.7) | 14.5 (2.7) | 14.6 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Who Experienced Ocular Anesthesia Following Treatment of AG-920 Compared to Placebo at 5 Minutes
Description: Immediately following EACH pinch test, subjects will be asked "Was that painful" "Yes" or "NO."
Time Frame: 5 minutes post dose
Measure: Count of Participants; unit: Participants
Arm/Group | AG-920 | Placebo
Number analyzed (Participants) | 60 | 60
Participants
  Anesthetic Response (painless) | 50 | 11
  No Anesthetic Response (pain) | 10 | 49

2. Secondary Outcome: How Long it Takes One Dose of AG-920 to Anesthetize the Eye
Description: Mean time to no pain score (onset)
Time Frame: 20, 40 and 60 seconds following dosing or until pain stops. 5-minutes post dose. If subject became anesthetized before 5 minutes, every 5 minutes for up to 30 minutes or until pain resumes.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | AG-920 | Placebo
Number analyzed (Participants) | 60 | 60
minutes | 0.43 (0.61) | 1.0 (1.67)

3. Secondary Outcome: How Long One Dose of AG-920 Anesthetizes the Eye
Description: Mean duration of anesthetic effect
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | AG-920 | Placebo
Number analyzed (Participants) | 60 | 60
minutes | 12.78 (7.97) | 6.61 (10.21)

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Total number of participants with TEAEs
Time Frame: from randomization through study completion (up to 5 days) on average of 2 days.
Measure: Count of Participants; unit: Participants
Arm/Group | AG-920 | Placebo
Number analyzed (Participants) | 60 | 60
Participants | 10 | 4

5. Secondary Outcome: Number of Participants With a Change in Biomicroscopy
Description: Slit lamp biomicroscopy and external eye exam measures will be summarized at each measured timepoint using discrete summary statistics. Clinician examined the eyelid, conjunctiva, cornea, anterior chamber, iris, pupil, and lens of the eye with the aid of a slit lamp.
Time Frame: change from baseline through end of study at Day 5
Population: Slit Lamp Examination Assessment change from baseline
Measure: Count of Participants; unit: Participants
Groups:
- AG-920: Articaine Sterile Topical Ophthalmic Solution (AG-920)
Arm/Group | AG-920 | Placebo
Number analyzed (Participants) | 60 | 60
Participants
  Study Eye | 0 | 0
  Fellow Eye | 0 | 0

6. Secondary Outcome: Change in Visual Acuity
Description: Visual Acuity data will be summarized at each time point using continuous and discrete summaries of Logarithmic Minimum Angle of Resolution (logMAR).
Time Frame: change from baseline through end of study at Day 5
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | AG-920 | Placebo
Number analyzed (Participants) | 60 | 60
LogMAR
  Study Eye | -0.03 (0.12) | -0.02 (0.06)
  Fellow Eye | -0.01 (0.05) | -0.02 (0.07)

ADVERSE EVENTS:
Time Frame: Adverse events were documented from the time the subject was consented until the subject's participation in the study was completed. This is a maximum of 6 days but an average of 2 days. If a subject had an ongoing AE at the time of study completion, the event was to be followed-up according to the site's standard of care and the subject provided appropriate medical care until the event resolved or stabilized.
Arm/Group | AG-920 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 7/60 | 2/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AG-920 (N=60) | Placebo (N=60)
conjunctival hyperemia (Eye disorders) | 7 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigative site, the Principal Investigator, and any other investigators understand and agree that the Study is a multi-center clinical study and that a multi-center publication may be prepared and published by the Sponsor. The investigative site and its investigators will not, individually or together, present or publish any findings, data or results of the Study.

DOCUMENTS (2):
  • Study Protocol (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT04829344/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT04829344/SAP_001.pdf